CLINICAL TRIAL: NCT03200873
Title: Effects of Repetitive Transcranial Magnetic Stimulation (rTMS) on Impulsivity and Empathy in a Non-clinical Population
Brief Title: Effects of rTMS on Impulsivity and Empathy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: C200317
Record Dates: First submitted 2017-06-13; First posted 2017-06-27 (Actual); Last update posted 2018-05-02 (Actual); Status verified 2017-10

CONDITIONS: Impulsive Behavior; Empathy
Keywords: transcranial magnetic stimulation; theta burst stimulation; impulsivity
MeSH Terms: conditions — Impulsive Behavior | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: crossover (real and sham stimulation) design with randomised allocation of outcome examination
Who Masked: Participant
Masking Description: using a shall coil to mimic the active stimulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- high impulsivity (Active Comparator): participants with high impulsivity (BIS >62), receiving active and sham repetitive transcranial magnetic stimulation [intermittent theta burst stimulation (iTBS)] in a randomised order
  Interventions: Device: repetitive transcranial magnetic stimulation
- low impulsivity (Active Comparator): participants with low impulsivity (BIS between 52 to 62), receiving active and sham repetitive transcranial magnetic stimulation [intermittent theta burst stimulation (iTBS)] in a randomised order
  Interventions: Device: repetitive transcranial magnetic stimulation

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — Each session of iTBS will apply3 trains of 600 pulses to the RDLPFC, with 20 2-second trains and an 8-second inter-train interval. Sham iTBS condition will be administered with the same methodology used for active iTBS condition with a sham coil mimicking noises and vibrations without delivery of magnetic pulses.
  Other Names: intermittent theta burst stimulation

SUMMARY:
Impulsivity describes the tendency to make risky and unplanned decisions, to pick immediate reward over a bigger reward after a period of time or to not be able to resist the urge to do something. Empathy refers to the ability to be sensitive to and vicariously experience other people's feelings and to create working models of emotional states. Recent neuroscientific research have found that the right frontal part of the brain (left dorsal lateral frontal cortex, LDLPFC) is important in the control of impulsive behaviour and empathy. Self-report questionnaires have been proven valid measures at assessing impulsivity and empathy. Repetitive Transcranial Magnetic Stimulation (rTMS) is a widely used non-invasive brain stimulation procedure; stimulation can be applied at different brain regions depending on the administration method. It temporally changes the way that this part of the brain functions, providing us a further understanding of how this part works. Recent research has found that rTMS on the LDLPFC changes performance-based tasks measuring different types of impulsivity and empathy. This study aims to investigate this further to look at the RDLPFC stimulation and its effects on empathy and two different types of impulsivity. Of interest is also how innate impulsive personality type and empathy trait relate to performance on these tasks.

DETAILED DESCRIPTION:
Background Impulsivity describes the tendency to make risky and unplanned decisions, to pick immediate reward over a bigger reward after a period or to not be able to resist the urge to do something. Empathy refers to the ability to be sensitive to and vicariously experience other people's feelings and to create working models of emotional states. Recent neuroscientific research have found that the left frontal part of the brain (left dorsal lateral frontal cortex, RDLPFC) is important in the control of impulsive behaviour and empathy. Self-report questionnaires have been proven valid measures at assessing impulsivity and empathy. Repetitive Transcranial Magnetic Stimulation (rTMS) is a widely used non-invasive brain stimulation procedure; stimulation can be applied at different brain regions depending on the administration method. It temporally changes the way that this part of the brain functions, providing us a further understanding of how this part works. Recent research has found that rTMS on the LDLPFC changes performance based tasks measuring different types of impulsivity and empathy. This study aims to investigate this further to look at the LDLPFC stimulation using the newer form of high-frequency rTMS, intermittent theta burst stimulation (iTBS) and its effects on empathy and two different types of impulsivity. Of interest is also how innate impulsive personality type and empathy trait relate to performance on these tasks.

Aims The specific purposes of this study are to (i) examine whether iTBS is an effective technique for modulating impulsivity and empathy, and to (ii) examine the relationship between the modulatory effects of the iTBS and baseline self-reported impulsivity and empathy.

The key objectives of this study are to examine whether the specific iTBS protocol at RDLPFC can effectively modulate two subtypes of impulsivity (delayed discounting and reflection impulsivity) and empathy, and to examine whether the participant's baseline self-reported impulsivity and empathy scores mediate the modulatory effects of the iTBS on impulsivity and empathy respectively in normal healthy young adults. The secondary objectives of this study are to examine whether the self-reported measures of impulsivity and empathy correlate with their performance-based counterparts.

Experimental protocol and methods The proposed study will be a single-centre, crossover design study, taking place at Queens Medical Centre, Nottinghamshire NHS Trust. Participants (male students or staff) will be recruited from the University of Nottingham. A potential participant will be asked to complete the TMS screening questionnaire to ensure that there are no contraindications to using TMS. After the written informed consent is obtained, he will then be asked to complete an online questionnaire (Barratt Impulsiveness Scale -version 11, BIS-11) measuring self-report impulsivity. The scores obtained from BIS-11 will be one of the screening criteria. If the potential participant is eligible for taking part in the study, he will be invited to the two laboratory sessions. He will then be asked to perform three computerised tasks assessing impulsivity and empathy before and after the iTBS administration. Each session of iTBS will apply 600 pulses to the LDLPFC, with 20 2-second trains and an 8-second inter-train interval for a total stimulation time of 190 seconds. Sham iTBS condition will be administered with the same methodology used for active iTBS condition with a sham coil mimicking noises and vibrations without delivery of magnetic pulses. Participants will be asked to guess which rTMS condition is real after completing the whole study to ascertain that whether the sham manipulation is successful or not. Participants will be monitored if they experience any adverse events during the rTMS session and instructed to report any experience of adverse events after each rTMS session. Tolerability will be presented as the number of reported adverse events and the number of dropouts due to adverse events.

Measurable end points/statistical power of the study To detect the change in impulsivity and empathy resulted from the iTBS intervention, G*Power 3.1.9.2 was used to estimate sample size required in consideration of interaction effect (impulsivity group × iTBS conditions) of repeated measure ANOVA. The following parameters were selected: effect size f = 0.20 (equivalent to d = 0.40, estimated from the results of previous meta-analyses), alpha error probability = .05, power = (1- β error probability) = .80, number of groups = 2, number of measurements = 2 and correlation among repeated measurements = 0.6. A minimum of total sample size of 42 subjects will be required. Considering the dropout rate of 0.20 (according to previous rTMS studies), 54 subjects will be required for the study, including 27 high impulsivity participants and 27 low impulsivity participants.

ELIGIBILITY:
Inclusion Criteria:

* Male students or staff in University of Nottingham
* aged 18-30 years.
* normal or corrected-to-normal vision
* BIS-11 scored above 71 or between 52 to 62
* Ability to give informed consent

Exclusion Criteria:

* Have ever suffered an epileptic fit
* Have had a brain injury or neurological disorder
* Have any non-removable metal implants in your head
* Have a family history of brain injury or epilepsy
* Drink more than 20 units of alcohol per week on a regular basis
* Currently take any illicit drugs
* Ever were dependent on illicit drugs or alcohol
* Ever suffered from a serious mental illness such as schizophrenia, severe depression or bipolar disorder
* Currently take any psychiatric medication

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males predominantly have higher impulsivity level compared to females
Enrollment: 33 (Actual)
Dates: Start 2017-05-17 (Actual); Primary Completion 2017-12-30 (Actual); Study Completion 2017-12-30 (Actual)

PRIMARY OUTCOMES:
Impulsivity (performance-based) | (usually 20 mins apart) the time just before rTMS and right after rTMS (usually 20 mins apart)
  P(correct) from IST and K value from AAT
empathy (performance-based) | baseline and right after rTMS (usually 20 mins apart)
  correct scores from RMET

SECONDARY OUTCOMES:
Correlation between self-reported and performance-based impulsivity | baseline
  correlation coefficient between [P(correct)], K value and AUC and UPPS-P and BIS-11
Correlation between self-reported and performance-based empathy | baseline
  correlation coefficient between RMET correct score and QCAE

OTHER OUTCOMES:
Incidence of Treatment-Emergent Adverse Events [Safety and Tolerability] | through study completion, an average within 1 week
  The frequency of adverse events from each participant

CONTACTS AND LOCATIONS:
Overall Officials: Birgit Völlm, PhD, Principal Investigator — Division of Psychiatry and Applied Psychology, School of Medicine, University of Nottingham
Locations (1):
- Division of Psychiatry and Applied Psychology, School of Medicine, University of Nottingham, Nottingham, Nottinghamshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No